CLINICAL TRIAL: NCT05532046
Title: A Phase 1b Double-blind, Randomized, Placebo-controlled, Multicenter, Dose Titration Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of 4 Weeks Treatment With BAY 2413555 in Participants With Heart Failure and Implanted Cardiac Defibrillator or Cardiac Resynchronization Devices
Brief Title: A Study to Learn How Safe Study Drug BAY2413555 is, How it Affects the Body, and How it Moves Into, Through, and Out of the Body Over 4 Weeks of Use in Participants With Heart Failure and Implanted Cardiac Defibrillator or Cardiac Resynchronization Devices (ICD/CRT)
Acronym: REMOTE-HF
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to new preclinical findings in a chronic toxicology study.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20623; 2021-005751-36 (EudraCT Number)
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment arm 1 (Experimental): Participants will receive BAY2413555 for 28 days (Part A: 14 days and Part B: 14 days).
  Interventions: Drug: BAY2413555 Dose 1
- Treatment arm 2 (Experimental): Participants will receive BAY2413555 for 28 days (Part A: 14 days and Part B: 14 days).
  Interventions: Drug: BAY2413555 Dose 1; Drug: BAY2413555 Dose 2
- Placebo (Placebo Comparator): Participants will receive placebo to BAY2413555 for 28 days (Part A: 14 days and Part B: 14 days).
  Interventions: Drug: Placebo to BAY2413555

INTERVENTIONS:
Drug: BAY2413555 Dose 1 — BAY2413555 Dose 1
  Arms: Treatment arm 1; Treatment arm 2
Drug: BAY2413555 Dose 2 — BAY2413555 Dose 2
  Arms: Treatment arm 2
Drug: Placebo to BAY2413555 — Placebo to BAY2413555
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat people who have chronic heart failure. Chronic heart failure is a medical condition with shortness of breath, tiredness and ankle swelling in which the heart does not pump blood as well as it should.

BAY2413555 is a new compound which is under development for the treatment of heart failure. Heart failure is a serious disease in which the heart pumps less well. BAY2413555 is expected to protect the heart and improve cardiac function.

The main purpose of this study is to learn how safe BAY2413555 is compared to placebo in participants with chronic heart failure and implanted cardiac defibrillator, or cardiac resynchronization devices (ICD/CRT). A placebo is a treatment that looks like a medicine, but does not have any medicine in it. ICD/CRT are machines placed in the body that use an electric shock/impulse to reset the heart or get it beating correctly. To study the safety, the researchers will record all medical problems the participants may have during the study after starting the study treatment. Medical problems that happen after the participants have started their treatment are also known as "treatment emergent adverse events" (TEAEs). The TEAEs will be compared between participants who received BAY2413555 and those who received placebo.

The second purpose of this study is to learn whether BAY2413555 effects electrical signals inside the heart compared to placebo.

The study has two parts, A and B. Each part will last for two weeks. In part A, the participants will be assigned by chance to either take BAY2413555 as a tablet by mouth once per day or a placebo. Participants from part A who do not need to stop the study based on predefined criteria continue in part B. They will be assigned by chance to receive either the same dose of BAY2413555 as in part A or a higher dose. Participants who have taken placebo in part A will as well be assigned in part B.

Each participant will be in the study for approximately 90 days (including the screening period and follow-up period). In the study, participants will take study medication for 28 days. 8 visits to the study site and 1 telephone contact visit are planned. During the study, the study team will:

* do physical examinations
* check vital signs
* examine heart health using ECG
* check the participants' ICD/CRT information
* take exercise testing
* take blood and urine samples
* ask the participants questions about how they are feeling about their quality of life
* ask the participants questions about how they are feeling and what adverse events they are having. An adverse event is any problem that happens during the trial. Doctors keep track of all adverse events that happen in trials, even if they do not think the adverse events might be related to the study treatments or a study procedure. Participants will be closely monitored during the entire study duration and site personnel will take action to mitigate any negative effect, if any, as appropriate.

About 30 days after the participants take their last treatment, the study doctors and their team will check the participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Providing signed informed consent
* Diagnosis of heart failure lasting for at least 3 months, New York Heart Association (NYHA) functional class I-III prior to Visit 1
* Left ventricular ejection fraction (LVEF) ≤ 45% as documented by any imaging modality within the past 12 months prior to Visit 1
* Treatment with Guideline-Directed Medical Therapy Including with mandatory betablocker treatment with either Metoprolol, Carvedilol, Bisoprolol or Nebivolol on stable, highest individually tolerated dose for at least 2 weeks prior to Visit 1
* Implanted cardiac defibrillator (ICD) with pacemaker backup function OR cardiac resynchronization device (CRT)

  * first implantation at least 3 months prior to Visit 1

Exclusion Criteria:

* Permanent atrial fibrillation or other than Sinus rhythm at Visit 1
* History of higher degree atrioventricular (AV) block (Mobitz type II or third-degree AV block) within 4 weeks prior to Visit 1
* Indication for or planned procedure:

  * Planned cardiac surgery, carotid angioplasty or surgery, transcatheter aortic valve implantation (TAVI) or mitral valve clipping within 3 months starting from the Screening Visit
  * Percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or implantation of a cardiac resynchronization therapy defibrillator device indicated at Screening or planned within 3 months starting from the Screening Visit
  * Valvular Disease Repair indicated at Screening or planned within 3 months starting from the Screening Visit.
* Occurrence of any of the following within 4 weeks prior to Visit 1:

  * Myocardial infarction
  * Stroke or transient ischemic attack (TIA)
  * coronary artery bypass graft (CABG)
  * percutaneous coronary intervention (PCI)
  * Carotid angioplasty
  * Ablation therapy of atrial fibrillation or other rhythm abnormalities
* Heart rate (HR) > 100 bpm at Screening Visit
* Restrictive, infiltrative or hypertrophic cardiomyopathy, constrictive pericarditis, acute myocarditis within 3 months prior to Visit 1
* Malignancy of the hematological system within 5 years prior to the Screening Visit
* Listed for heart transplantation and/or anticipated implantation of a ventricular assist device at the Screening Visit
* Hepatic insufficiency classified as Child-Pugh B or C at the Screening Visit
* Estimated (according to the investigator's judgement) inability to perform exercise testing
* Any of the following from the blood sample taken at the Screening Visit

  * Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2 (calculated according to the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation)
  * Hemoglobin < 11 g/dL
  * White blood cell (WBC) < 3000/mm^3
  * Thrombocytes < 100 000/mm^3
* Currently receiving or planned to receive dialysis or ultrafiltration
* Chronic obstructive pulmonary disease (COPD) Stage 3 or 4 (GOLD criteria), requiring treatment, or symptomatic asthma requiring current treatment
* Prior or concomitant therapy with cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors or inducers.

Relevant substances need to be discontinued

* at least 2 weeks before randomization for CYP3A4 inducers
* at least 5 half-lives before randomization for CYP3A4 inhibitors Restarting of these therapies is possible 28 days after last intake of study intervention. This criterion also applies to other inhibitors of CYP3A4, e.g., grapefruit.

Prior and concomitant therapy with amiodarone is allowed.

* Concomitant treatment with acetylcholine esterase inhibitors within 4 weeks prior to Visit 1
* Use of other investigational drugs. Previous (within 4 weeks, or 5 half-lives of the investigational drug, whichever is longer, prior to Visit 1) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s)
* Life expectancy < 6 months at the Screening Visit

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 56 days

SECONDARY OUTCOMES:
Number of participants with higher degree atrioventricular (AV) blocks, symptomatic pauses/bradycardia | Up to 28 days
Changes from baseline in resting heart rate (HR) after 2 and 4 weeks of dosing with BAY2413555 | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (18):
- United States (3):
  - Accel Research Sites - Atlanta Clinical Research Center, Atlanta, Georgia
  - White Oak Medical Center, Silver Spring, Maryland
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
- Denmark (3):
  - Capital Region | Gentofte Hospital - Cardiology Research, Hellerup
  - Odense Universitetshospital, Hjertemedicinsk Amb., Odense C
  - Zealand University Hospital | Roskilde - Cardiology Department, Roskilde
- Pratia | Klinische Forschung Dresden, Dresden, Saxony, Germany
- Israel (3):
  - Barzilai Ashkelon University Medical Center | Cardiology Department, Ashkelon
  - Rambam Health Care Campus | Internal Medicine - Cardiology Department, Haifa
  - Ziv Medical Center | Cardiology Department, Safed
- Italy (2):
  - Humanitas Research Hospital | Cardio Center - Clinical, Interventional Cardiology and Coronary Care, Milan, Lombardy
  - Fondazione Toscana Gabriele Monasterio | Heart Hospital Gaetano Pasquinucci - Cardiology Department, Pisa, Tuscany
- Spain (6):
  - Hospital Alvaro Cunqueiro | Cardiology Department, Babio - Beade, Pontevedra
  - Hospital del Mar | Cardiology Department, Barcelona
  - Hospital Universitari de Bellvitge | Bellvitge Biomedical Research Institute - Cardiology Department, Barcelona
  - Junta de Andalucía | University Hospital Reina Sofia - Cardiology Department, Córdoba
  - Hospital Universitario Virgen de la Victoria | Cardiology Department, Málaga
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/20623